CLINICAL TRIAL: NCT06722846
Title: Communicating Health Options to Inform Care and Empower Strategic Care Planning (CHOICES): A Multi-layer Randomized Case Vignette Study.
Status: Recruiting | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2024-0531; NCI-2024-10042 (Other: NCI-CTRP Clinical Registry)
Record Dates: First submitted 2024-12-03; First posted 2024-12-09 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Health Options; Strategic Care Planning

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Randomized Case Vignette Study: If participants agree to take part in this study, participants will complete about 16 questionnaires that will have questions about participants quality of life, anxiety, health, and case scenarios that are not real or based on your actual health situation. It should take a bit more than an hour to complete all the questionnaires. If participants find that any of these questions are difficult to read, understand, or otherwise complete; or if they cause distress, participants may ask the study team for clarification, skip the question, or even stop the study at any time.
  Additionally, information will be collected from participants medical record about participants health and treatment, as well as participants demographic information (age, race, sex, and so on). Investigators may also ask participants for additional demographic information not found in your medical record.
  Interventions: Behavioral: Randomized Case Vignette Study

INTERVENTIONS:
Behavioral: Randomized Case Vignette Study — Particpants will complete about 16 questionnaires that will have questions about particpants quality of life, anxiety, health, andcase scenarios that are not real or based on particpants actual health situation.

SUMMARY:
To learn more about how the delivery of medical information affects therapy choices for participants with advanced forms of cancer.

DETAILED DESCRIPTION:
Primary Objectives • To examine how provision of medical information (risks, benefits, time toxicity, prognosis, oncologists' recommendation, and costs) affects preference for palliative systemic therapy in participants with advanced cancer.

Secondary Objective

• To examine how different options of medical information (risks/benefits, time toxicity, prognosis, oncologists' recommendation, and costs) affect preference for palliative systemic therapy in participants with advanced cancer.

Exploratory Objective

* To examine how the order of presentation of medical information affects preference for palliative systemic therapy in participants with advanced cancer.
* To examine the association between intrinsic participants characteristics (such as participants demographics, symptoms, anxiety, depression, illness understanding, acceptance, coping strategies, religious coping, hope, decision making style, trust in oncologist, financial distress) and preference for palliative systemic therapy in participants with advanced cancer.

ELIGIBILITY:
Inclusion Criteria:

Diagnosis of advanced solid tumor (i.e. metastatic, relapsed, and/or incurable disease) or aggressive lymphoma.

* Age 18 or greater
* Seen at MD Anderson Cancer Center Thoracic and Lymphoma Oncology Clinics for a follow-up visit
* Been treated with at least 2 lines of palliative systemic cancer therapies

Exclusion Criteria:

* Diagnosis of cognitive impairment or dementia requiring a surrogate decision maker
* Non-English speaking

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: MD Anderson Cancer Center
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2024-11-21 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2028-08-31 (Estimated)

PRIMARY OUTCOMES:
Overall Survival (OS) | Through study completion; an average of 1 year.
  Progression Free Survival (PFS)

CONTACTS AND LOCATIONS:
Overall Officials: David Hui, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org

DOCUMENTS (1):
  • Informed Consent Form (2024-11-07): https://cdn.clinicaltrials.gov/large-docs/46/NCT06722846/ICF_000.pdf